CLINICAL TRIAL: NCT06228248
Title: Characterizing the Differences in Gut Microbiome Antibiotics Resistance Gene Between Healthcare Workers and the Healthy Population
Brief Title: Antibiotics Resistance Gene in Healthcare Workers
Acronym: ARGH
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Lingtong Huang, MD, Principal investigator, First Affiliated Hospital of Zhejiang University
Other Study IDs: IIT20230455B
Record Dates: First submitted 2024-01-02; First posted 2024-01-29 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2024-02

CONDITIONS: Multidrug Resistant Bacterial Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Fecal specimens are used for extracting DNA and conducting metagenomic sequencing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- medical worker: Medical workers working in clinical settings, including nurses, doctors, and Health care worker.
  Interventions: Other: metagenomics
- health population: Healthy individuals who do not engage in medical work
  Interventions: Other: metagenomics

INTERVENTIONS:
Other: metagenomics — Feces used for metagenomic testing

SUMMARY:
Multidrug resistant bacteria (MDR) pose a threat to the safety of patients worldwide. Drug resistant bacteria are commonly present in hospital environments and can cause infections, often leading to outbreaks within hospitals. Cross transmission through medical staff has been proven to be a significant cause of MDR bacterial transmission in hospitals. Although some studies have shown that the detection of gut drug-resistant bacteria in healthcare workers is similar to that in healthy individuals, these studies are limited to small sample sizes and detection methods. Here, the investigator characterize the differences between ARG colonization among healthcare workers and healthy populations through deep metagenomics.

DETAILED DESCRIPTION:
Understanding the antibiotic resistant genes in the intestinal microbiome of medical workers can reveal their exposure history to antibiotics and the status of antibiotic resistance. The gut microbiome of medical staff may be one of the important sources of MDR transmission. The contact between medical staff and patients is one of the main ways of MDR transmission in hospitals. Understanding the types and distribution of antibiotic resistant genes of gut microbiome of medical workers can assess the risk of MDR transmission in the hospital, help to assess them as the potential source of MDR transmission, and then take targeted prevention and control measures.

In order to better understand the role of medical staff in the transmission of MDR, it is necessary to conduct research on larger sample size and more sensitive detection methods. Metagenomics studies the genomes of all microorganisms in the microbial ecological community. It constructs a metagenomic library by directly extracting the DNA or RNA of all microorganisms from environmental samples, studies the species composition and functional composition of the community, the interaction of different microorganisms in the same population, and the interaction between microbial communities and hosts, and makes a comparative analysis of samples with different phenotypes. With the characteristics of high data flux, low cost and fast speed, it has become a powerful tool for the study of gut microbe.

To sum up, MDR poses a serious threat to global security. In order to deal with this problem, more in-depth and comprehensive research is needed to understand the transmission route of MDR in the hospital. The investigator evaluated the difference between the gut microbe antibiotic resistant genes abundance of medical workers, especially medical workers in the ICU, and healthy people through in-depth sequencing, which helps to provide information on the potential role of medical staff in the transmission of MDR, and is essential for formulating effective prevention and control strategies.

ELIGIBILITY:
For medical workers:

Inclusion Criteria:

1. Age greater than 18 years old
2. The subjects fully understand and sign the informed consent form

Exclusion Criteria:

1. Existence of gastrointestinal diseases, malignant tumors, and psychiatric disorders
2. Have taken broad-spectrum antibiotics within 6 months
3. Pregnant women

For healthy control:

Inclusion Criteria:

1. Age greater than 18 years old
2. The subjects fully understand and sign the informed consent form

Exclusion Criteria:

1. Previously or currently engaged in medical related work
2. Existence of gastrointestinal diseases, malignant tumors, and psychiatric disorders
3. Have taken broad-spectrum antibiotics within 6 months
4. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study included medical workers and health control. The investigator excluded underlying diseases that may have an impact on the gut microbiome, and also excluded individuals who had used broad-spectrum antibiotics within 6 months.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-11-10 (Actual)

PRIMARY OUTCOMES:
Differences in GUT ARG abundance between two groups | 1 year
  After conducting metagenomic testing, the investigator will analyze the raw data according to the preset protocol process and report the gut ARG abundance of different individuals. Subsequently, the difference in ARG abundance between the two groups of patients will be compared.

SECONDARY OUTCOMES:
The association of occupational exposure time in the ICU environment and ARG | 1 year
  After conducting metagenomic testing, the investigator will analyze the raw data according to the preset protocol process and report the gut ARG abundance of different individuals. Subsequently, the investigator will assess the correlation between occupational exposure time in the ICU environment and ARGs abundance of two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Lingtong Huang, M.D., Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (8):
- China (8):
  - First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Hospital of Jiaxing, Jiaxing
  - Lishui People's Hospital, Lishui
  - The First People's Hospital of Pinghu, Pinghu
  - Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University, Taizhou
  - Henan Provincial People's Hospital, Zhengzhou
  - The Fifth Clinical Medical College of Henan University of Chinese Medicine, Zhengzhou
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: Undecided
Contact Dr. Lingtong Huang to obtain IPD data

REFERENCES:
- [Derived] Huang L, Li K, Peng C, Gu S, Huang X, Gao C, Ren X, Cheng M, He G, Xu Y, Jiang Y, Wang H, Wang M, Shen P, Wang Q, He X, Zhong L, Wang S, Wang N, Zhang G, Cai H, Jiang C. Elevated antibiotic resistance gene abundance of ICU healthcare workers, a multicentre, cross-sectional study. Crit Care. 2025 Apr 30;29(1):170. doi: 10.1186/s13054-025-05408-5. PMID 40307838